CLINICAL TRIAL: NCT00926224
Title: Fibroscan® and Its Dedicated Probes Efficiency in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Responsible Party: Celine Fournier, Echosens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M111
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Liver Fibrosis; Cirrhosis
Keywords: Adult patients with chronic liver disease scheduled for a liver biopsy and a BMI superior or equal to 28 kg/m²
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

INTERVENTIONS:
Device: FibroScan M and XL probes — Each patient undergo two liver stiffness measurements with the FibroScan: once with the M probe and once with the XL probe

SUMMARY:
The main objective of the study is to evaluate the diagnostic performance of the XL probe for estimating degree of liver fibrosis/cirrhosis in obese patients > 28 kg/m² with various liver diseases in patients with chronic liver disease scheduled for a liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient of at least 18 years of age
* Patient able to give written informed consent form
* Patient with a BMI superior or equal to 28kg/m²
* Patient scheduled to have a liver biopsy within 1 month after the enrollment or with a liver biopsy performed within 6 months before the enrollment.
* Patient for which abdominal ultrasound is technically possible

Exclusion Criteria:

* Unable or unwilling to provide written informed consent
* Confirmed diagnosis and/or history of malignancy, or other terminal disease
* Patients with clinical ascites
* Pregnant women
* Patient with a BMI < 28 kg/m²
* Patients with any active implantable medical device (such as pacemaker or defibrillator)
* Transplanted patient and patient with heart disease
* Refusal to undergo a liver biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
diagnosis accuracy for the assement of significant fibrosis and cirrhosis | at enrollement

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Calgary University Hospital, Calgary, Alberta
  - London University Hospital, London, Ontario
  - Toronto Western General Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Saint-Luc University, Montreal, Quebec